CLINICAL TRIAL: NCT02267174
Title: Handoffs and Transitions in Critical Care (HATRICC): Optimizing Operating Room to Intensive Care Unit Handoffs
Brief Title: Handoffs and Transitions in Critical Care
Acronym: HATRICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Anesthesia Patient Safety Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AWD-10044739, 819726
Record Dates: First submitted 2014-10-07; First posted 2014-10-17 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Patient Handoff; Healthcare Team; Communication; Patient Safety; Intensive Care Units
Keywords: Implementation; quality improvement; patient safety; handoffs; intensive care unit; postoperative care; simulation
MeSH Terms: conditions — Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standardized OR to ICU handoff (Other): A standardized handoff process for conducting OR to ICU handoffs will be implemented in two intensive care units without a standard process.
  Interventions: Behavioral: Standardized handoff

INTERVENTIONS:
Behavioral: Standardized handoff — A standardized handoff will be implemented that consists of choreographed handoffs utilizing a structured handoff tool to facilitate information exchange.

SUMMARY:
The HATRICC study will use mixed methods to implement a standardized process for operating room to intensive care unit handoffs that is accepted and sustainably used by perioperative clinicians.

DETAILED DESCRIPTION:
BACKGROUND: Operating room to intensive care unit handoffs are high-risk events for critically ill patients. Studies in selected patient populations show that standardizing operating room to intensive care unit handoffs improves information exchange and decreases errors. To adapt these findings to mixed surgical populations, the investigators propose to study the implementation of a standardized operating room to intensive care unit handoff process in two intensive care units currently without an existing standard process. METHODS/DESIGN: The Handoffs and Transitions in Critical Care (HATRICC) study is a hybrid effectiveness-implementation trial of operating room to intensive care unit handoffs. The investigators will use mixed methods to conduct a needs assessment of the current handoff process, adapt published handoff processes, and implement a new standardized handoff process in two academic intensive care units. Needs assessment - The investigators will use nonparticipant observation to observe the current handoff process. Focus groups, interviews, and surveys of clinicians will elicit participants' impressions about the current process. Adaptation and implementation - The investigators will adapt published standardized handoff processes using the needs assessment findings. The investigators will use small group simulation to test the new process' feasibility. After simulation, the investigators will incorporate the new handoff process into the clinical work of all providers in the study units. Evaluation - Using the same methods employed in the needs assessment phase, the investigators will evaluate use of the new handoff process. Data analysis - The primary effectiveness outcome is the number of information omissions per handoff episode as compared to the pre-intervention period. Additional intervention outcomes include patient intensive care unit length of stay and intensive care unit mortality. The primary implementation outcome is acceptability of the new process. Additional implementation outcomes include feasibility, fidelity and sustainability. DISCUSSION: The HATRICC study will examine the effectiveness and implementation of a standardized operating room to intensive care unit handoff process. Findings from this study have the potential to improve healthcare communication and outcomes for critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* All clinicians caring for patients being transferred from the operating room to intensive care unit.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in information omissions | baseline to 1 month post-intervention
  The number of information omissions per handoff episodes will be determined by direct observation.

SECONDARY OUTCOMES:
Change in teamwork score | baseline to 1 month post-intervention
  Quantitative teamwork score will be determined for each episode of operating room to intensive care unit handoff after the intervention is implemented.
Change in patient length of stay | baseline to 1 month post-intervention
  Patient length of stay in the intensive care unit and in the hospital will be assessed in the post-intervention period.

OTHER OUTCOMES:
Change in qualitative implementation outcomes | baseline to 1 month post-intervention
  Acceptability, appropriateness and fidelity will be assessed qualitatively

CONTACTS AND LOCATIONS:
Overall Officials: Meghan B Lane-Fall, MD, MSHP, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lane-Fall MB, Pascual JL, Peifer HG, Di Taranti LJ, Collard ML, Jablonski J, Gutsche JT, Halpern SD, Barg FK, Fleisher LA; HATRICC study team (Kimberly Allen, BSN, RN; Mark Barry, MD; Sruthi Buddai, BA; Tyler Chavez, BA; Mahrukh Choudhary, BA; Della George; Megan Linehan, DO; Enrique Torres Hernandez; Jerome Watts, BA. A Partially Structured Postoperative Handoff Protocol Improves Communication in 2 Mixed Surgical Intensive Care Units: Findings From the Handoffs and Transitions in Critical Care (HATRICC) Prospective Cohort Study. Ann Surg. 2020 Mar;271(3):484-493. doi: 10.1097/SLA.0000000000003137. PMID 30499797
- [Derived] Lane-Fall MB, Beidas RS, Pascual JL, Collard ML, Peifer HG, Chavez TJ, Barry ME, Gutsche JT, Halpern SD, Fleisher LA, Barg FK. Handoffs and transitions in critical care (HATRICC): protocol for a mixed methods study of operating room to intensive care unit handoffs. BMC Surg. 2014 Nov 19;14:96. doi: 10.1186/1471-2482-14-96. PMID 25410548
- See also: Study website — http://www.hatricc.com